CLINICAL TRIAL: NCT06445478
Title: Comparison of Blood Flow Restrictive Exercises and Isokinetic Exercises in Female Football Players: Randomized Controlled Study
Brief Title: Effectiveness of Blood Flow Restricting Exercises and Isokinetic Exercises in Female Football Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, Ebru Sever, Lecturer, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: İREMNURESMANURRABİA
Record Dates: First submitted 2024-04-29; First posted 2024-06-06 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Female Football Players
Keywords: Resistance exercise; Isokinetic exercise; Female football player; Blood flow restrictive exercise; Athlete rehabilitation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Resistant exercise with blood flow restrictive exercise (BFR-RE Group )) (Experimental): Resistant exercise with blood flow restrictive exercise (BFR-RE) training will be given 2 days a week for 8 weeks. Each exercise session will consist of 4 sets. There will be 30 repetitions in the first set and 15 repetitions in the next 3 sets, for a total of 75 repetitions. There will be a minimum of 30 seconds and a maximum of 60 seconds of rest intervals between sets. Since the application will be performed for the lower extremity muscle groups, a cuff will be placed on the proximal part of the lower extremity. Exercise load will be determined as 20-40% of 1 RM.
  Interventions: Other: Blood Flow Restrictive Exercise and Isokinetic Exercise
- Group 2 (Resistant exercise with isokinetic device (ID-RE Group)) (Experimental): Resistant exercise with isokinetic device (ID-RE) training will be given 2 days a week for 8 weeks. During the training, leg press, squat and knee extension movements will be improved by increasing the resistance or changing the position depending on the athlete's condition.
  Interventions: Other: Blood Flow Restrictive Exercise and Isokinetic Exercise

INTERVENTIONS:
Other: Blood Flow Restrictive Exercise and Isokinetic Exercise — Before providing exercise training, the muscle strength, circumference measurement, joint range of motion, agility and quality of life of female football players will be determined. Muscle strength measurements will be evaluated with the Kineo Intelligent Load Isokinetic Device for the BFR-RE and ID-RE groups. Then, both groups will be given 4 weeks of resistance exercise training. After this training, all evaluations will be made again. After this evaluation, another 4 weeks of training will be given and the evaluations will be re-applied at the end of the 8th week.
  The "Informed Volunteer Consent Form" will be read and signed by 30 selected participants.

SUMMARY:
Our aim in the study is; Comparison of blood flow restrictive exercises and isokinetic exercises in female football players. 30 female football players between the ages of 18-30 who came to DOIT Health & Sports clinic to receive rehabilitation will be included in the study. Participants will be randomized into 2 groups. Resistant exercise with blood flow restrictive exercise (BFR-RE) will be applied to one group, and resistant exercise with isokinetic device (ID-RE) will be applied to the other group. An 8-week exercise protocol will be created for both groups and exercise training will be given twice a week. Demographic data form, Kineo Intelligent Load Isokinetic Device to measure muscle strength, tape measure to measure circumference, universal goniometer for joint range of motion, Illinois Agility Test for agility and quality of life; World Health Organization Quality of Life Scale-Short Form Turkish Version will be administered before exercise, at the 4th week and at the 8th week. The effectiveness of the applications for female football players and their advantages over each other will be examined. The 4-week and 8-week effects of 2 types of exercise will be examined.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-30
* Becoming a female football player
* Volunteering to participate in the study

Exclusion Criteria:

* Deep vein thrombosis
* Pregnancy
* Hypertension
* Anti-inflammatory use
* Unexplained chest pain
* Congenital heart disease
* Participants with a history of contraindications to exercise
* There is another study conducted at the same time as the study.

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-04-02 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Kineo Intelligent Load Isokinetic Device | 10 weeks
  With Kineo, evaluation of lower/upper extremity and trunk muscles can be made. The device can also be used to provide strength training. The isokinetic method is characterized by movement at a predetermined constant speed regardless of the applied force. The test (single or double-sided) includes 5 consecutive movements with different speed and maximum power connection. Analysis of the graph allows evaluation of the relationship between force, velocity and angle. It allows isokinetic exercise to be performed at all workstations, both in the open chain and in the closed chain. Additionally, with Kineo Biphasic Load, it is possible to distinguish the load between concentric and eccentric phases to reduce muscle effort and make the work safer. Detailed reports on strength, muscle imbalances and all data necessary for continuous monitoring of the rehabilitation process are instantly visible, can be printed or exported in Excel format.
Thigh and Leg Circumference Measurement | 10 weeks
  A foldable, non-elastic 7 mm wide tape measure will be used for circumference measurements. The tape measure will not be affected by the tensions during the measurement and the "0" starting part will be in the left hand, the area to be measured with the other hand will be wrapped with the tape measure and the circumference will be measured by placing the "0" point and the measured number side by side rather than on top of each other.
Universal Goniometer | 10 weeks
  Flexion and extension range of motion (ROM) of the knee was measured in degrees (°) using the "Universal Goniometer". Knee ROM was assessed using a goniometer with the participant lying supine with the heel elevated on a foam roller. Knee extension was measured with participants maximally extending the knee joint and was defined as the difference from 0° extension. Knee flexion was measured with patients bending their knees and lifting their heels toward their hips as far as possible. The pivot point of the goniometer was placed on the lateral condyle of the femur, and the fixed arm was placed on the lateral side of the leg in the direction of the midline of the femur, and the measurement was made so that the movable arm followed the movement of the fibula.
Illinois Agility Test | 10 weeks
  It is used to determine the agility of athletes by taking into account their direction changes. Before the test, necessary explanations are made and the track is introduced, then the subjects are allowed to make 3-4 attempts at a low tempo. It is performed on a test track consisting of three cones arranged in a straight line with a width of 5 m, a length of 10 m and 3.3 m intervals in the middle section. The test consists of a slalom run, with 180° turns every 10 m, 40 m on the flat and 20 m between cones. Athletes are asked to start at the starting line of the test track, lying face down and with their hands in contact with the ground at shoulder level. With complete rest, the test is repeated 2 times and the best value is recorded in seconds.
World Health Organization Quality of Life Scale - Short Form Turkish Version | 10 weeks
  The health-related quality of life scale was developed by WHO, and its validity and reliability were tested by Eser et al. The scale has two versions: long (WHOQOL-100) and short (WHOQOL-27) form. The scale measures physical, spiritual, social and environmental well-being and consists of 26 questions. The scale can be applied to non-elderly adults. Since each domain expresses the quality of life in its own field independently of each other, domain scores are calculated between 4-20. As the score increases, the quality of life increases.

CONTACTS AND LOCATIONS:
Locations (1):
- DOIT Health & Sports Clinic, Istanbul, Ataşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No